CLINICAL TRIAL: NCT01676233
Title: A Randomized, Open-label, 2-treatment Crossover Study of a New Formulation of Insulin Glargine Comparing to Lantus® on 24-hour Glucose Profile in Japanese Patients With Type 1 Diabetes Mellitus on Treatment With Basal-bolus Insulin
Brief Title: Repeated Dose Study With a New Insulin Glargine Formulation and Lantus® on 24-hour Glucose Profile in Japanese Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDY12335; U1111-1129-3633 (Other: UTN)
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Reference (insulin glargine) -Test1 (insulin glargine - new formulation), both dose will be adjusted individually to achieve the target glycemic goal
  Interventions: Drug: insulin glargine (HOE901); Drug: insulin glargine- new formulation (HOE901)
- Sequence 2 (Experimental): Test1 - Reference , both dose will be adjusted individually to achieve the target glycemic goal
  Interventions: Drug: insulin glargine (HOE901); Drug: insulin glargine- new formulation (HOE901)

INTERVENTIONS:
Drug: insulin glargine (HOE901) — Pharmaceutical form: solution Route of administration: subcutaneous
Drug: insulin glargine- new formulation (HOE901) — Pharmaceutical form: solution Route of administration: subcutaneous

SUMMARY:
Primary Objective:

- To compare the 24-hour glycemic profile in continuous glucose monitoring (CGM) between a new formulation of insulin glargine and Lantus at steady state

Secondary Objectives:

* To compare the change of Fasting plasma glucose (FPG), Self-monitoring plasma glucose (SMPG) and Postprandial Plasma Glucose (PPG) between the 2 treatments;
* To compare the efficacy of the 2 treatments on glycemic control in glycemic parameters (1,5-anhydroglucitol and hemoglobin A1c (glycosylated hemoglobin; HbA1c));
* To compare the occurrence of hypoglycemia between the 2 treatments;
* To assess the safety and tolerability of a new formulation of insulin glargine.

DETAILED DESCRIPTION:
66 days

ELIGIBILITY:
Inclusion criteria :

* Japanese patients with Type 1 Diabetes Mellitus (T1DM) on treatment with basal-bolus insulin;

Exclusion criteria:

* Age < 20 years at written informed consent;
* HbA1c < 6.5% or > 10.0% at screening
* Diabetes mellitus (DM) other than T1DM;
* Body Mass Index (BMI) > 35.0 kg/m2 at screening visit
* Any contraindication to use of insulin glargine as defined in the Japanese Package Insert
* Hypoglycemia unawareness or history of metabolic acidosis, including hospitalization for diabetic ketoacidosis during the 24 weeks prior to screening visit

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour blood glucose profile measured by continuous glucose monitoring | Baseline, Day 28, Day 56

SECONDARY OUTCOMES:
Hypoglycemia categorized by the definition of American Diabetes Association | Up to Day 56
Change in fasting plasma glucose from baseline to each treatment end by treatment | Baseline, Day 28, Day 56
Change in self monitoring plasma glucose profile from baseline to each treatment end by treatment | Baseline, Day 28, Day 56
Change in HbA1c from baseline to each treatment end by treatment | Baseline, Day 28, Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 392001, Kumamoto, Japan

REFERENCES:
- [Derived] Jinnouchi H, Koyama M, Amano A, Takahashi Y, Yoshida A, Hieshima K, Sugiyama S, Kurinami N, Jinnouchi T, Becker R. Continuous Glucose Monitoring During Basal-Bolus Therapy Using Insulin Glargine 300 U mL(-1) and Glargine 100 U mL (-1) in Japanese People with Type 1 Diabetes Mellitus: A Crossover Pilot Study. Diabetes Ther. 2015 Jun;6(2):143-52. doi: 10.1007/s13300-015-0115-1. Epub 2015 Jun 9. PMID 26055218